CLINICAL TRIAL: NCT06275503
Title: STROKESTOP III - Optimized Method for Atrial Fibrillation Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); Landstinget i Värmland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STROKESTOP III
Record Dates: First submitted 2023-11-06; First posted 2024-02-23 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation New Onset
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic screening group (Other): Individuals aged 75/76 randomized to systematic screening are invited through a centralized screening facility to participate in prolonged ECG screening.
  Interventions: Behavioral: Screening invitation mode
- Opportunistic screening group (Other): Individuals aged 75/76 randomized to opportunistic screening are invited to participate when they visit their primary care facility to prolonged ECG screening.
  Interventions: Behavioral: Screening invitation mode

INTERVENTIONS:
Behavioral: Screening invitation mode — Cluster randomized study to compare mode of invitation

SUMMARY:
Atrial fibrillation is the most common sustained cardiac arrhythmia affecting more than 3% of the adult population. The symptoms of atrial fibrillation can range from asymptomatic to debilitating. It can be permanent in its nature, but also paroxysmal with only short bursts of atrial fibrillation randomly occurring and can therefore remain unnoticed. Atrial fibrillation increases the risk of stroke five fold if left untreated.

Screening for atrial fibrillation in elderly populations above age 65 years can result in detection of new atrial fibrillation cases ranging from 0,5% new AF with a single time-point ECG, up to 30% AF if an implantable loop recorder is inserted for 3 years.

Currently opportunistic screening using pulse palpation, or a single time-point ECG is recommended by the European Society of Cardiology guidelines. Systematic screening in individuals aged 75 or above, or at a high stroke risk should be considered.

Overall, participation in systematic atrial fibrillation screening trials has been shown to be relatively low with almost 50% non-participants. Participants are generally healthier, with higher socioeconomic status, hence the ones who would potentially benefit the most remain absent.

Opportunistic screening has shown promising results with higher participation rates and the possibility of better outreach. There is a lack of data from randomized trials on the difference in participation rates in systematic and opportunistic screening approaches when screening with prolonged ECG monitoring.

DETAILED DESCRIPTION:
Plans and methods; Primary care facilities in the region of Värmland with at least 200 75-76 year-old listed will be randomized to either:

1. Systematic screening. All 75/76 year old belonging to a primary care facility randomized to systematic screening will receive a letter with an invitation to screening through the Clinical Physiology department at Karlstad Central Hospital.
2. Opportunistic screening. All 75/76 year old attending their primary care facility for any health related reason will be invited to screening at the primary care facility.

A complete list of all listed individuals will be drawn from each primary care facility list of patients for both screening arms at the beginning of the study.

Inclusion criteria: All individuals aged 75/76 residing in the region of Värmland, listed at a primary care facility with > 200 individuals aged 75/76 Exclusion criteria: Individuals with ongoing oral anti coagulation treatment (OAC), contraindication for OAC treatment and/or known and treated atrial fibrillation will be excluded from participation. Individuals not being able to consent will be excluded from participation.

All participants will be asked to fill out a health declaration. A hand-held single-lead ECG (Zenicor One) will be sent to the participant via mail. The device will be used to measure ECGs on a regular basis three times a day, and during symptoms. ECGs are transferred for interpretation through the mobile network. All ECGs will be manually interpreted by specifically trained physiologists.

All positive findings are communicated to primary care by the physiologists for initiation of OAC treatment. All negative findings are communicated to the participant via mail.

Participation status, and new AF diagnosis will be assessed immediately after study closure. Secondary endpoints will be assessed at one year through Swedish national patients' registries.

In a sub-study an artificial intelligence model will be scoring all individuals' risk of developing AF based on the initial ECG (unless there is substantial noise, then second ECG will be used). The AI analysis will be blinded to the interpreter of the ECGs. All participants will be stratified into a low-risk and a high-risk group of developing AF during screening based on the AI analysis. At the end of the screening period the outcome of the AI model will be compared with the results of the screening.

In a sub study the investigators will use artificial intelligence as a means of assessment support when interpreting ECGs. The artificial intelligence model has been used to determine a cut-off for high and low risk individuals and will be prospectively evaluated to determine if it can be used to identify individuals that will benefit most from AF screening.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 75/76 in 2024 (born 1948, 1949)
* Must reside in the region of Värmland
* Must be listed at a primary care facility

Exclusion Criteria:

* Treatment with oral anti coagulation treatment (OAC)
* Contraindications for OAC treatment
* Prior atrial fibrillation
* Unable to provide consent

Ages: 75 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Participation in screening | 12 months
  Proportion of invitees participating in screening in each screening arm. The primary hypothesis is that opportunistic screening will increase participation by 25 % compared to systematic screening

SECONDARY OUTCOMES:
AF detection in opportunistic compared to systematic screening | 12 months
  Proportion of participants with newly diagnosed AF in the screening groups
OAC treatment after AF detection | 12 months
  Proportion of participants with AF on OAC treatment after AF detection by manual follow up
Compliance to OAC treatment 1 year after initiation | 12 months
  Proportion of participants with AF on OAC treatment after AF detection
Health economy | 12 months
  Health-economic assessment of costs accrued in the systematic screening group compared to the opportunistic screening group
Composite endpoint of stroke, death and severe bleeding | 5 years
  A combined endpoint of the rate of stroke, all-cause death and severe bleeding leading to hospitalization in the group randomized to systematic screening compared to opportunistic screening
Reminder strategy effect on participation | 12 months
  The proportional increase in participation after reminder letter is sent out in both groups.
Comparison of automatic ECG analysis (using AI) for detection of AF in a (by AI algorithm classified) high- compared to a low-risk group | 12 months
  Proportion of new AF detected in the group determined as high risk per AI-algorithm compared to the group marked as low risk by the AI algorithm.
  An AI-algorithm using a neural network has previously been developed (PMID: 36881777) and will be prospectively tested to determine if individuals classified as high-risk to develop AF by the AI-algorithm on their initial electrocardiogram have an increased risk of screening-detected AF. The ECG reviewers will be blinded to the result of the AI-algorithm.
Application of the FIND-AF algorithm | 12 months
  An artificial intelligence model developed from electronic health care records in the United Kingdom has shown an increased risk of incident atrial fibrillation. We aim to determine how accurate the pre-specified variables from the FIND-AF algorithm (age, gender, presence of valvular disease, chronic pulmonary disease, chronic renal failure, as well as Chads-Vasc parameters) can predict atrial fibrillation (reported by sensitivity, specificity and area under the curve).

CONTACTS AND LOCATIONS:
Overall Officials: Emma Svennberg, MD PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Dept Med H, Stockholm
  - Region Värmland, Värmland

IPD SHARING:
Plan to Share IPD: No